CLINICAL TRIAL: NCT06607289
Title: National Longitudinal Cohort of Hematological Diseases (NICHE) - CART
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2024047
Record Dates: First submitted 2024-09-01; First posted 2024-09-23 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-09

CONDITIONS: Hematological Malignancies
Keywords: Chimeric antigen receptors (CAR) T cell; hematological malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, ambispective, longitudinal, observational cohort study investigating CAR-T cell therapy in Chinese patients with hematological malignancies. A consortium of Phase IV clinical trials and real-world studies of Chimeric antigen receptors (CAR) T cell therapy will be established in China. Patient-level data from these studies will be collected to create a large real-world cohort. In addition, patients receiving CAR-T cell therapy for hematological malignancies identified from an existing hematology longitudinal cohort study, the National Longitudinal Cohort of Hematological Diseases (NICHE), will also be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed hematologic malignancies
* Patients treated with CAR-T cell therapy
* Signed the informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematologic malignancies treated with Chimeric antigen receptors (CAR) T therapy in China
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term overall remission rate | 5 years
  Proportion of the participants with an overall remission. To investigate the long-term efficacy of Chimeric antigen receptors (CAR) T cell therapy in Chinese patients with various hematological malignancies.

SECONDARY OUTCOMES:
Complete remission rate | 1 year, 2 years, 5 years
  Proportion of the participants with an complete remission. To investigate the long-term efficacy of Chimeric antigen receptors (CAR) T cell therapy in Chinese patients with various hematological malignancies.
Partial remission rate | 1 year, 2 years, 5 years
  Proportion of the participants with an partial remission. To investigate the long-term efficacy of Chimeric antigen receptors (CAR) T cell therapy in Chinese patients with various hematological malignancies.
Long-term safety | 5 years or more
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
  To investigate the long-term safety of Chimeric antigen receptors (CAR) T cell therapy in Chinese patients with various hematological malignancies.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China